CLINICAL TRIAL: NCT01726829
Title: Overnight Type 1 Diabetes Control Under MD-Logic Closed Loop System at the Patient's Home, Pilot Study.
Brief Title: Overnight Type 1 Diabetes Control Under MD-Logic Closed Loop System at the Patient's Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: rmc007053ctil
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Artificial Pancreas; Closed Loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MD-Logic Artificial Pancreas (MDLAP) system (Experimental): four consecutive outpatients overnight sessions at home under closed loop MD-Logic Artificial Pancreas (MDLAP) system
  Interventions: Device: MD-Logic Artificial Pancreas (MDLAP) system
- Standard treatment with sensor augmented pump therapy (Active Comparator): four consecutive outpatients overnight sessions at home under standard treatment with sensor augmented pump therapy
  Interventions: Procedure: sensor augmented pump therapy

INTERVENTIONS:
Device: MD-Logic Artificial Pancreas (MDLAP) system
  Other Names: four consecutive outpatients overnight sessions at home under closed loop MD-Logic Artificial Pancreas (MDLAP) system
  Arms: MD-Logic Artificial Pancreas (MDLAP) system
Procedure: sensor augmented pump therapy
  Other Names: four consecutive outpatients overnight sessions at home under standard treatment with sensor augmented pump therapy
  Arms: Standard treatment with sensor augmented pump therapy

SUMMARY:
This is a randomized prospective single blind trial to evaluate blood glucose control overnight under closed-loop insulin delivery with MD-Logic Artificial Pancreas (MDLAP) system in patients with type 1 diabetes, being conducted in: Tel Aviv, Israel, Ljubljana, Slovenia and Hannover, Germany; In this study,75 eligible patients will be enrolled.Each subject will participate in four consecutive over nights under closed-loop with MDLAP, and four additional over nights under regular sensor augmented pump therapy at home with a washout period of 10 ± 3 days between arms.

DETAILED DESCRIPTION:
In the last two decades, remarkable technological progress has been made with the development of continuous glucose sensors, miniature devices, implantable pumps and sensors and wireless communications, interest in the closed-loop insulin delivery was revived.

Control trails that evaluate the clinical benefits of continuous glucose sensor have shown improved HbA1c with no significant increase in sever hypoglycemia, trend towards lower hypoglycemic episodes although not significant and no significant change in sever hypoglycemia. One of the main drawbacks of continuous glucose sensor is noncompliant of the patient, the flow of information and the need to act accordingly makes this devise a burden for some patients. Theoretically subcutaneous insulin pumps and glucose sensors attached to an artificial pancreas in a closed-loop system can mimic the activity of functioning pancreatic beta cells, with strict control of blood glucose levels. Such a system may also offer an opportunity to free the patients from the daily burden of dealing with their diabetes.

Study Objectives are to determine the safety and efficacy of using the MDLAP system to automatically control overnight blood glucose in type 1 diabetic patients. Overnight glucose control time defined as the time range between bedtime (21:00-23:00 PM) and awaking time (7:00 AM).

This is a randomized prospective single blind trial to evaluate blood glucose control overnight under closed-loop insulin delivery with MD-Logic Artificial Pancreas (MDLAP) system in patients with type 1 diabetes, being conducted in: Tel Aviv, Israel, Ljubljana, Slovenia and Hannover, Germany; 75 eligible patients will be enrolled.Each subject will participate in four consecutive over nights under closed-loop with MDLAP, and four additional over nights under regular sensor augmented pump therapy at home with a washout period of 10 ± 3 days between arms.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 diabetes (>1yr since diagnosis)
* Insulin infusion pump therapy for at least 3 months
* Patients whom used continuous glucose sensor previously
* Age at inclusion ≥ 10 years and ≤ 65 years
* HbA1c at inclusion ≥ 7 and <10
* Patients willing to follow study instructions
* Patients live with at least one other adult person
* BMI SDS(Standard Deviation Score) - below the 97th percentile for age
* An internet connection at patient's home
* Patients with care givers who are capable of operating a computer based system

Exclusion Criteria:

* Concomitant diseases that influence metabolic control
* Participation in any other interventional study
* Known or suspected allergy to trial products
* Any significant diseases (such as preexisting seizures or epilepsy) or conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subjects ability to complete the study or compromise patients safety
* Diabetic ketoacidosis in the past 1 month
* Severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrollment.
* Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Female subject who is pregnant or planning to become pregnant within the planned study duration

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
time sensor glucose level spent below 70mg/dl | final visit (day 44)
The percentage of nights mean overnight sensor glucose levels was within90-140 mg/dl | At final visit (day 44)

SECONDARY OUTCOMES:
The time sensor glucose level spent within 70-140 mg/dl | At final visit (day 44)
The number and frequency of hypoglycemic events below 63, 79 mg/dl | At final visit (day 44)
The time sensor glucose level spent above 140, 180 mg/dl | At final visit (day 44)
The area under the curve <63, <70, >140, >180 mg/dl | At final visit (day 44)
Glucose variability | At final visit (day 44)
  glucose variability measured as the standard deviation from the mean glucose
The total insulin dose during the overnight period | At the final visit (day 44)
Artificial pancreas technical performance defined as total frequency of technical failures | at final visit (day 44)
Artificial pancreas technical performance defined as total frequency of lost or inaccurate sensor records | At final vist (day 44)
Percentage of time of active closed loop control | At final visit (day 44)
  percentage of time that the MDLAP system worked without any technical problem
Fear of Hypoglycemia questionnaire | At final visit (day 44)
Acceptance questionnaire | At final visit (day 44)
Artificial Pancreas Satisfaction Questionnaire | At final visit (day 44)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, MD, Principal Investigator — Schneider Children's Medical Center
Locations (3):
- Diabetes -Zentrum fuer kinder und jugendliche, Hanover, Germany
- Schneider Children's Medical Center, Petah Tikva, Israel
- University Children's Hospital, Slovenia, Slovenia

REFERENCES:
- [Derived] Nimri R, Muller I, Atlas E, Miller S, Kordonouri O, Bratina N, Tsioli C, Stefanija MA, Danne T, Battelino T, Phillip M. Night glucose control with MD-Logic artificial pancreas in home setting: a single blind, randomized crossover trial-interim analysis. Pediatr Diabetes. 2014 Mar;15(2):91-9. doi: 10.1111/pedi.12071. Epub 2013 Aug 15. PMID 23944875